CLINICAL TRIAL: NCT02377947
Title: A Retrospective, Open-label, Uncontrolled Cohort Study to Assess the Effectiveness and Safety of Lactulose Retention Enema in the Treatment of Cirrhotic Patients With Grade 3 or 4 (West Haven Criteria) Hepatic Encephalopathy (HE) [The RETRO Study]
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: EPIDJ001; REF/2014/11/007981 (Registry Identifier: Clinical Trial registry of India)
Record Dates: First submitted 2015-02-17; First posted 2015-03-04 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Hepatic Encephalopathy
Keywords: Lactulose Retention Enema; Hepatic Encephalopathy, Grade 3 or 4 West Haven Criteria; The Retro Study
MeSH Terms: conditions — Hepatic Encephalopathy; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with cirrhosis (grade 3 & 4 per west haven cr.): Patients with cirrhosis having grade 3 or grade 4 (West Haven Criteria) hepatic encephalopathy who were treated with Lactulose retention enema

SUMMARY:
This is a retrospective study in adult patients with cirrhosis and grade 3 or 4 HE (West Haven Criteria) to evaluate the effectiveness and safety of lactulose retention enema in the treatment of deep grade HE (West Haven Criteria). The study will be conducted retrospectively in a multi center of a multispecialty tertiary care hospital in India, in which lactulose retention enema is the mainstay of management of cirrhotic patients with grade 3 or 4 HE (West Haven criteria). Dosing of lactulose retention enema in this study will be done according to the dosing described for rectal administration of lactulose (India): 300ml of lactulose mixed with 700ml of potable water to be used as a retention enema; the enema is to be retained for 30-60 minutes and repeated every 4-6 hours until the patient is able to take oral medication. This treatment regime is also the standard protocol of management of deep grade HE (West Haven criteria) in the study centers. The standard treatment protocol of deep grade HE (West Haven criteria) of the study centers will also ensure that all known contraindications of lactulose will be respected before administration of lactulose retention enema to the study patients. The retrospective hospital records of the patient population of interest within the past 6 months will be identified, and these records will be used to collect data required for analysis.

DETAILED DESCRIPTION:
Data to be collected:

Data that would be collected for the study as part of retrospective chart review:

1. Patient demographics: age, gender, weight
2. Medical history
3. Etiology of cirrhosis (alcohol abuse, hepatitis, autoimmune, cryptogenic, other)
4. Diagnosis of cirrhosis
5. History of previous HE (if yes, the number of episodes in the past)
6. Grade of HE (as per the West-Haven criteria) at admission, 24 hrs and 48 hours post treatment with lactulose
7. Precipitating factor(s) of HE (Dehydration, GI bleeding, protein overload, constipation, infection, others)
8. Dose and duration of lactulose enema
9. Treatment given for precipitating factors
10. Laboratory data on haemoglobin, platelet, bilirubin, albumin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), urea, creatinine, sodium, potassium, and blood ammonia
11. Complete reversal of deep-grade HE (< Grade 2 as per West-Haven criteria) (yes/no)
12. Time to complete reversal of deep-grade HE
13. Number of days in hospital
14. Adverse drug reaction experienced by the patient
15. Complications experienced by the patient
16. Other pharmacovigilance relevant information (OPRI)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years of either gender.
* Patients admitted to the hospital with liver cirrhosis and grade 3 or grade 4 (West Haven Criteria) HE
* Patients treated with lactulose retention enema within 48 hours of onset of grade 3 or 4 (West Haven Criteria) HE

Exclusion Criteria:

* Patients treated with agents other than lactulose retention enema for grade 3 or 4 (West Haven Criteria) HE.
* Patients who had significant concomitant diseases that could impair or contribute to the impairment of consciousness
* Patients who had a major neuropsychiatric illness
* Patients who had a contraindication to lactulose, including Hypersensitivity to the active substance or to any of the ingredients; Galactosaemia; Gastrointestinal obstruction, digestive perforation or risk of digestive perforation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective study - data charts of the cirrhotic patients having grade III and IV and who were administered lactulose enema will be reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dyotona Roy-Sengupta, Study Chair — Abbott
Locations (3):
- India (3):
  - Medanta Hospital, Gūrgaon
  - Research facility ORG-000333, Gūrgaon
  - Sir Ganga Ram Hospital, New Delhi

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Cirrhosis (Grade 3 & 4 Per West Haven cr.)
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Cirrhosis (Grade 3 & 4 Per West Haven cr.)
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.38 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 40
Region of Enrollment [Count of Participants; unit: Participants]
  India | 50

OUTCOME MEASURES:

1. Primary Outcome: Complete Reversal
Description: Percentage of patients with complete reversal of deep-grade (Grade 3 and 4 West-Haven Criteria) Hepatic Encephalopathy after administration of lactulose retention enema
Time Frame: 24 hrs
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Patients With Cirrhosis (Grade 3 & 4 Per West Haven cr.)
Number analyzed (Participants) | 50
percentage of participants | 80 [66.3 to 90.0]

2. Primary Outcome: Complete Reversal
Description: as for outcome 1
Time Frame: 48 hrs
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Patients With Cirrhosis (Grade 3 & 4 Per West Haven cr.)
Number analyzed (Participants) | 50
percentage of participants | 90 [78.2 to 96.7]

3. Secondary Outcome: Hepatic Encephalopathy (HE) Grade Shift at 24 and 48 Hours
Description: Grade shift at 24 and 48 hours - from baseline to 24 and 48 hours post administration of lactulose retention enema.
  Complete reversal of deep grade HE is defined as subjects having HE grade=<grade 2 as per West-Haven criteria where grade 0 is Normal, Grade 1 is Mild lack of awareness, Grade 2 is Lethargic, Grade 3 is Somnolent but arousable and Grade 4 is Coma
Time Frame: HE Grade shift at 24 hrs and HE Grade shift at 48 hrs
Measure: Number; unit: percentage of participants
Arm/Group | Patients With Cirrhosis (Grade 3 & 4 Per West Haven cr.)
Number analyzed (Participants) | 50
percentage of participants
  shift from HE Grade 3 to <2 after 24 hours | 86.67
  shift from HE Grade 4 to <2 after 24 hours | 20.0
  shift from HE Grade 3 to <2 after 48 hours | 95.56
  shift from HE Grade 4 to <2 after 48 hours | 40.0

4. Secondary Outcome: Time to Complete Reversal
Description: Time to complete reversal of deep-grade (Grade 3 and 4 West-Haven Criteria) HE after administration of lactulose retention enema
Time Frame: up to 48 hrs
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Patients With Cirrhosis (Grade 3 & 4 Per West Haven cr.)
Number analyzed (Participants) | 50
Hours | 25.39 (8.85)

5. Secondary Outcome: Mortality
Description: Mortality in patients treated with lactulose retention enema
Time Frame: within 48 hrs
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Cirrhosis (Grade 3 & 4 Per West Haven cr.)
Number analyzed (Participants) | 50
Participants | 0

6. Other Pre Specified Outcome: Safety of Lactulose Retention Enema (Number of Adverse Drug Reactions & Complications).
Description: Safety of Lactulose retention enema (number of adverse drug reactions & complications). Complications pertinent to lactulose retention enema are in reference to potential adverse effects associated with the use of rectal device associated with the application of the lactulose retention enema kit.
Time Frame: Chart Review of Events over 48 Hour Period
Measure: Number; unit: number of events
Arm/Group | Patients With Cirrhosis (Grade 3 & 4 Per West Haven cr.)
Number analyzed (Participants) | 50
number of events | 5

7. Other Pre Specified Outcome: Reduction in Blood Ammonia Level
Description: Change from baseline was calculated at the end of treatment by using following formula wherever applicable:
  Change from baseline = Blood ammonia level at the end of treatment - Blood ammonia level at baseline
Time Frame: reported at 48 hrs
Population: The ammonia levels were available at baseline for 28 patients where as the last observed blood ammonia level after administration of lactulose enema was available for 4 patients. Thus the change from baseline was calculated for 4 patients. The Change value = Visit value - Baseline Value
Measure: Mean (Standard Deviation); unit: Mcg/DL
Arm/Group | Patients With Cirrhosis (Grade 3 & 4 Per West Haven cr.)
Number analyzed (Participants) | 4
Mcg/DL | -70.6 (11.32)

8. Other Pre Specified Outcome: Duration of Hospital Stay
Time Frame: upto 30 days of hospital admission
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Patients With Cirrhosis (Grade 3 & 4 Per West Haven cr.)
Number analyzed (Participants) | 50
hours | 229.4 (147.64)

ADVERSE EVENTS:
Description: As this study was a retrospective chart review of 50 patients who were treated with lactulose enema, only (S)ADRs and complications were collected. Thus, the total of participants at risk were 50 for ADRs and complications. Complications pertinent to lactulose retention enema are in reference to potential adverse effects associated with the use of rectal device associated with the application of the lactulose retention enema kit.
Arm/Group | Patients With Cirrhosis (Grade 3 & 4 Per West Haven cr.)
All-Cause Mortality (participants affected / at risk) | 6/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 3/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Cirrhosis (Grade 3 & 4 Per West Haven cr.) (N=50)
Diarrhea and Abdominal discomfort (Gastrointestinal disorders) | 1 (2) — Only ADRs and complications were collected. Observed non serious ADRs are either considered to be sufficiently described in the section on undesirable effects in local label and/or associated with the method of administration as a retention enema
Abdominal fullness and discomfort (Gastrointestinal disorders) | 1 (2) — Only ADRs and complications were collected. Observed non serious ADRs are either considered to be sufficiently described in the section on undesirable effects in local label and/or associated with the method of administration as a retention enema
Mild rectal bleed (Injury, poisoning and procedural complications) | 1 (1) — Only ADRs and complications were collected. Observed non serious ADRs are either considered to be sufficiently described in the section on undesirable effects in local label and/or associated with the method of administration as a retention enema

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No